CLINICAL TRIAL: NCT00162058
Title: An Open-Label, Non-Randomized, Phase II Trial To Assess Focal Liver Lesion Detection Using Definity-Enhanced Ultrasound Imaging
Brief Title: A Phase II Study of DMP 115 to Assess Focal Liver Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Qi Zhu, MD Sr. Medical Director, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DMP 115-214
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

INTERVENTIONS:
Drug: Peflutren Lipid Microsphere Injectable Suspension

SUMMARY:
To determine the optimal dose of DMP 115 to image liver lesions and to assess whether contrast can improve the detection of focal liver lesions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with 1 but <7 focal liver lesions
* Scheduled for liver biopsy within 30 days of study
* Scheduled for CT or MR within 30 days of study

Exclusion Criteria:

* Critically ill subjects
* Subjects with right-to-left shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The ratio of signal intensities obtained from unenhanced vs. contrast-enhanced ultrasound imaging of liver tissue and liver lesions will be calculated at the end of the study.

SECONDARY OUTCOMES:
The determination of the presence or absence of focal liver lesions during the Blinded Read and the Institutional Read of ultrasound images.

CONTACTS AND LOCATIONS:
Overall Officials: Edward L.S. Leen, MD, Principal Investigator — Consultant Radiologist, Royal Infirmary
Locations (1):
- Local Institution, Glasgow, Scotland, United Kingdom